CLINICAL TRIAL: NCT00608933
Title: CAM USE and Cancer
Brief Title: Education Intervention in Encouraging Health Providers to Talk With Cancer Patients About the Use of Complementary and Alternative Medicine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2006-0198; MDA-2006-0198; NCI Clinical Trials (Other: CDR0000584715); 5U10CA045809-17 (NIH); NCI-2009-00005 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-01-30; First posted 2008-02-06 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Arm I (intervention) (Active Comparator): Health providers receive educational materials comprising a brief video about communicating with and providing guidance to patients regarding complimentary and alternative medicine (CAM) and a list of resources they can access to obtain information about herbs, CAM modalities, and drug/herb interactions. Approximately 2 weeks after the educational intervention, health providers receive a follow-up e-mail reminding them to ask patients about CAM use. The e-mail also includes a brief update regarding current research findings on CAM modalities and drug/herb interactions.
  Interventions: Other: educational intervention; Other: questionnaire administration
- Arm II (wait-list) (Other): Health providers are enrolled on a wait-list. After 2 months, the educational materials in arm I (educational intervention) are made available to the wait-list health providers.
  Interventions: Other: educational intervention; Other: questionnaire administration

INTERVENTIONS:
Other: educational intervention — Health providers receive educational materials comprising a brief video about communicating with and providing guidance to patients regarding complimentary and alternative medicine (CAM) and a list of resources they can access to obtain information about herbs, CAM modalities, and drug/herb interactions. Approximately 2 weeks after the educational intervention, health providers receive a follow-up e-mail reminding them to ask patients about CAM use. The e-mail also includes a brief update regarding current research findings on CAM modalities and drug/herb interactions.
Other: questionnaire administration — Patients complete questionnaires

SUMMARY:
RATIONALE: Educating health providers on talking with cancer patients about complementary and alternative medicine (CAM) may help encourage health providers to talk more often with cancer patients about the use of CAM.

PURPOSE: This randomized phase III trial is studying how well an education intervention works in encouraging health providers to talk with cancer patients about the use of CAM.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Examine the efficacy of an education intervention designed to increase the frequency with which health providers ask cancer patients about their use of complimentary and alternative medicine (CAM).

Secondary

* Examine the frequency with which health providers ask about CAM use and referral for CAM use by health providers.
* Evaluate whether personal CAM use among health providers is related to the frequency of asking patients about CAM use.
* Assess the frequency and type of CAM use among patients diagnosed with cancer.

OUTLINE: This is a multicenter study. Stratification is based on the number of health providers at each CCOP component site (< 3 health providers per component site vs 3 to 6 health providers per component site vs 7 to 9 health providers per component site vs 10 or more health providers per component site). The CCOP component sites are randomized to 1 of 2 intervention groups.

* Arm I (intervention): Health providers receive educational materials comprising a brief video about communicating with and providing guidance to patients regarding complimentary and alternative medicine (CAM) and a list of resources they can access to obtain information about herbs, CAM modalities, and drug/herb interactions. Approximately 2 weeks after the educational intervention, health providers receive a follow-up e-mail reminding them to ask patients about CAM use. The e-mail also includes a brief update regarding current research findings on CAM modalities and drug/herb interactions.
* Arm II (wait-list): Health providers are enrolled on a wait-list. After 2 months, the educational materials in arm I are made available to the wait-list health providers.

Health providers in both arms complete questionnaires at baseline and at 2 months to assess the effectiveness of the educational intervention, personal CAM use, and level of knowledge about CAM and to determine if they are asking patients about CAM use. Patients of the health providers also complete questionnaires at the same time points to assess personal CAM use before and after cancer diagnosis as well as the level of their interaction with health providers regarding CAM use.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Health provider meeting the following criteria:

  * Has regular contact with cancer patients by initially talking with patients, taking their histories, and conveying pertinent information to their physician at a participating CCOP site

    * Must be actively seeing patients at a participating University of Texas (UT) MD Anderson Cancer Center Community Clinical Oncology Program (CCOP) site
  * Must not be employed at more than one participating CCOP site
  * Not a temporary employee
* Patient of a health provider at a participating CCOP site meeting the following criteria:

  * Current diagnosis of cancer including amyloidosis

    * Diagnosed at least 1 week ago
    * Finished treatment within the past 6 months
  * Able to speak or read English
  * No prior participation in this study at an earlier assessment

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1356 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who report that the health provider discussed complimentary and alternative medicine (CAM) use | Baseline to 2 months
  The Complementary and Alternative Medicine Patient Survey administered to patients to assess personal use of CAM before and after the cancer diagnosis as well as the level of interaction with providers regarding CAM use. Baseline survey assessment at one week and follow up assessment at 2 months.

SECONDARY OUTCOMES:
Frequency with which health providers ask about CAM use and referral for CAM use by health providers | Baseline to 2 months
Relationship between personal CAM use among health providers and frequency of asking patients about CAM use | Baseline to 2 months
Frequency and type of CAM use among patients diagnosed with cancer | Up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas